CLINICAL TRIAL: NCT06867913
Title: A Pilot Study of Selenomethionine and Myo-inositol(SOLOWAYS_TM) in Patients With Autoimmune Thyroiditis Carrying the DIO2 Thr92Ala Polymorphism
Brief Title: A Study of Selenomethionine and Myo-inositol(SOLOWAYS_TM) in Patients With Autoimmune Thyroiditis Carrying the DIO2 Thr92Ala Polymorphism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Collaborators: Center for New Medical Technologies, Novosibirsk, Russia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SW022
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Autoimmune Thyroiditis
Keywords: Thyroid gland; genetics; supplements; anti-TPO; T4; T3
MeSH Terms: conditions — Thyroiditis, Autoimmune; Thyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Thr92Ala Carriers) (Experimental)
  Interventions: Dietary Supplement: Supplement groupx
- Cohort B (Wild-Type DIO2) (Experimental)
  Interventions: Dietary Supplement: Supplement groupx

INTERVENTIONS:
Dietary Supplement: Supplement groupx — Selenomethionine (e.g., 100 µg/day)
  * Myo-inositol (e.g., 600 mg/day or higher)
  * Patients on levothyroxine will maintain their current dose (if clinically indicated).
  Arms: Cohort A (Thr92Ala Carriers)
Dietary Supplement: Supplement groupx — Selenomethionine (e.g., 100 µg/day)
  * Myo-inositol (e.g., 600 mg/day or higher)
  * Patients on levothyroxine will maintain their current dose (if clinically indicated).
  Arms: Cohort B (Wild-Type DIO2)

SUMMARY:
This pilot, genotype-stratified clinical trial aims to evaluate the safety and preliminary efficacy of combined selenomethionine and myo-inositol supplementation in patients with autoimmune thyroiditis (AIT), including Hashimoto's thyroiditis, who carry the Thr92Ala (rs225014) variant in the DIO2 gene. The study will compare changes in thyroid function tests, autoantibody titers, and clinical symptoms between two cohorts: (1) carriers (homozygous or heterozygous) of the Thr92Ala variant and (2) individuals without this variant ("wild-type"). The hypothesis is that patients with the "unfavorable" DIO2 genotype will experience greater improvements in TSH levels, the free T3/ free T4 ratio, and autoimmunity markers when receiving selenomethionine plus myo-inositol, potentially due to enhanced support of thyroid hormone conversion and reduced autoimmune activity.

DETAILED DESCRIPTION:
Rationale

* The DIO2 gene encodes the type II iodothyronine deiodinase, which converts T4 (thyroxine) to the more active T3 (triiodothyronine) in peripheral tissues.
* The Thr92Ala (rs225014) polymorphism may reduce enzyme activity, potentially leading to lower tissue T3 levels, even in patients with normal or slightly elevated T4 and TSH.
* Selenium (as selenomethionine) supports the function of various selenoproteins, including deiodinases, and has been reported to reduce anti-thyroid antibody levels (particularly anti-TPO).
* Myo-inositol has shown promise in modulating autoimmune and metabolic processes in thyroid disorders, possibly improving tissue sensitivity to thyroid hormones and reducing autoimmune inflammation.
* A genotype-focused approach may reveal whether individuals carrying the DIO2 Thr92Ala variant derive a more substantial benefit from combined supplementation than those without the variant. 2. Study Goals
* Primary Goal: To assess changes in TSH levels and the fT3/fT4 ratio over 12 weeks of combined selenomethionine and myo-inositol supplementation.
* Secondary Goals:

  * To evaluate changes in thyroid autoantibody titers (anti-TPO, anti-Tg).
  * To assess thyroid ultrasound findings (vascularization, gland volume).
  * To measure improvements in patient-reported symptoms and quality of life using standardized questionnaires.
  * To determine the safety and tolerability of the combined intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years with a clinical diagnosis of autoimmune thyroiditis (elevated anti- TPO and/or anti-Tg).
* TSH range consistent with subclinical hypothyroidism (e.g., TSH 4.5-10 mIU/L) or euthyroid status with AIT; patients on stable levothyroxine therapy are eligible if dose was unchanged for at least 6 weeks.
* Willingness to undergo genotyping for the DIO2 Thr92Ala variant. Confirmation of the Thr92Ala variant (homozygous or heterozygous) for Cohort A; absence of this variant for Cohort B.
* Ability to provide informed consent and comply with study procedures.

Exclusion Criteria:

* Overt hypothyroidism with TSH >10 mIU/L requiring immediate treatment adjustment.
* Significant comorbidities (e.g., uncompensated heart failure, severe renal or hepatic dysfunction, uncontrolled diabetes).
* Pregnancy or lactation (given potential changes in thyroid requirements and supplement safety considerations).
* Known hypersensitivity to selenium or inositol supplements.
* Severe psychiatric disorder interfering with protocol adherence.
* Concurrent use of high-dose selenium (>50 µg/day) or other thyroid-influencing nutraceuticals that cannot be discontinued prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-12-26 (Actual); Study Completion 2025-02-21 (Actual)

PRIMARY OUTCOMES:
Change in Serum Thyroid-Stimulating Hormone (TSH) Concentration | 16 weeks
  Change in serum TSH concentration (reported in µIU/mL) from baseline to 16 weeks. The results will be presented as the mean change in concentration.
Change in Serum Free T3/Free T4 Ratio | 16 weeks
  Change in the ratio of serum free triiodothyronine (fT3) to free thyroxine (fT4) from baseline to 16 weeks. The outcome will be reported as the mean ratio change.

SECONDARY OUTCOMES:
Change in Serum Anti-Thyroid Peroxidase (anti-TPO) Antibody Concentration | 16 weeks
  Change in the concentration of serum anti-thyroid peroxidase (anti-TPO) antibodies (measured in IU/mL) from baseline to 16 weeks. The outcome will be reported as the mean change in antibody concentration.
Change in Serum Anti-Thyroglobulin (anti-Tg) Antibody Concentration | 16 weeks
  Change in the concentration of serum anti-thyroglobulin (anti-Tg) antibodies (measured in IU/mL) from baseline to 16 weeks. The outcome will be reported as the mean change in antibody concentration.
Thyroid Gland Ultrasound Measurements: Volume | 12 weeks
  Ultrasound assessment of the thyroid gland will include measurement of thyroid volume (in mL) and qualitative assessment of thyroid echogenicity. Thyroid volume will be calculated using standardized ultrasound techniques, and echogenicity will be rated using a predetermined grading system.
Change in Patient-Reported Symptom Severity | 12 weeks
  Patient-reported symptom severity will be assessed using the Patient Health Questionnaire-15 [PHQ-15]). , if the PHQ-15, scores range from 0 to 30, with higher scores indicating worse symptom severity. The outcome will be reported as the mean change in symptom severity score from baseline to 12 weeks.
Number of incidence of any Treatment-Related Adverse Events | 12 weeks
  The incidence of treatment-related adverse events will be recorded and graded using the Common Terminology Criteria for Adverse Events (CTCAE v4.0). Data will be reported as the number and percentage of participants experiencing one or more adverse events.
Change in Patient-Reported Quality of Life | 12 weeks
  Quality of life will be assessed using a validated instrument such as the World Health Organization Quality of Life-BREF (WHOQOL-BREF). For instance, scores for each domain range from 0 to 100, with higher scores indicating a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No